CLINICAL TRIAL: NCT04105335
Title: An Open Label Phase 1a/b Study of MTL-CEBPA in Combination With a PD-1 Inhibitor (Pembrolizumab) in Adult Patients With Advanced Solid Tumours
Brief Title: A Study of MTL-CEBPA in Combination With a PD-1 Inhibitor in Patients With Advanced Solid Tumours (TIMEPOINT)
Acronym: TIMEPOINT
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mina Alpha Limited (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: MNA-3521-012; 2019-002231-28 (EudraCT Number)
Record Dates: First submitted 2019-08-16; First posted 2019-09-26 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2023-06

CONDITIONS: Solid Tumor, Adult
Keywords: Oligonucleotide; saRNA; Pembrolizumab; Tumour microenvironment; Myeloid-derived suppressor cells; C/EBP-a; CEBPA
MeSH Terms: interventions — pembrolizumab

STUDY DESIGN:
Intervention Model Description: The principal objective of the first part of the study (Phase 1a) is to establish if a combination of an experimental drug (MTL-CEBPA) with pembrolizumab (PD-1 inhibitor) is safe and well-tolerated in patients with advanced solid tumours.
  Phase 1b will aim to confirm the doses of the drugs obtained in Phase 1a in a larger population and if it has potential to reduce the size of the tumour and/or extend the life of participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Cohort 1 MTL-CEBPA in combination with pembrolizumab (Experimental): MTL-CEBPA 70mg/m2 administered weekly over 3 weeks followed by 1 week of rest combined with pembrolizumab 200mg administered every 3 weeks.
  Interventions: Drug: MTL-CEBPA; Drug: Pembrolizumab
- Cohort 2 MTL-CEBPA in combination with pembrolizumab (Experimental): MTL-CEBPA 98mg/m2 administered weekly over 3 weeks followed by 1 week of rest combined with pembrolizumab 200mg administered every 3 weeks.
  Interventions: Drug: MTL-CEBPA; Drug: Pembrolizumab
- Cohort 3 MTL-CEBPA in combination with pembrolizumab (Experimental): MTL-CEBPA 130mg/m2 administered weekly over 3 weeks followed by 1 week of rest combined with pembrolizumab 200mg administered every 3 weeks.
  Interventions: Drug: MTL-CEBPA; Drug: Pembrolizumab
- Expansion Cohort MTL-CEBPA in combination with pembrolizumab (Experimental): MTL-CEBPA RP2D administered once every 3 weeks on Day 1 of every 3 week cycle. Pembrolizumab 200mg administered once 3 weeks on Day 8 of every 3 week cycle.
  Interventions: Drug: MTL-CEBPA; Drug: Pembrolizumab

INTERVENTIONS:
Drug: MTL-CEBPA — Intravenous administration
Drug: Pembrolizumab — Intravenous administration
  Other Names: Keytruda

SUMMARY:
This is an open label Phase 1a/1b study in patients who have advanced solid cancer tumours. Patients will receive MTL-CEBPA (an experimental drug) in combination with pembrolizumab (a drug which has been given approval for use for some tumour types).

The Phase 1a dose escalation part of the study is designed to establish which doses of MTL-CEBPA are safe and well-tolerated when combined with the standard dose of pembrolizumab. Patients recruited to this part of the study will be those whose cancer progressed on standard treatment(s) or for whom no treatments are available.

Phase 1b the dose expansion part of the study will further explore how safe and well-tolerated these two drugs are when combined and will assess if the combination of drugs could potentially reduce the size of tumours. Participants in this part of the study will receive the experimental drug (MTL-CEBPA) at a dose which is considered safe and well-tolerated based on data from the first part of the study (Phase 1a). Participants will remain in the study taking study drugs until either death, or they choose to withdraw from the study.

DETAILED DESCRIPTION:
Phase 1a comprises three planned dose cohorts (ascending dose, 3+3 design, at the following dose levels: 70 mg/m2 QW, 98 mg/m2 QW, and 130 mg/m2 QW) of MTL-CEBPA combined with standard dose of pembrolizumab (given every 3 weeks). The aim is to assess the safety and tolerability of MTL-CEBPA in combination with pembrolizumab, recruiting patients whose disease progressed on standard of care therapy or for whom no therapy is available.

In the first dose cohort the first participant enrolled will receive MTL-CEBPA treatment at the 70mg/m2 QW dose level. Pembrolizumab (200mg) will be administered on Day 2 of the first cycle and subsequently every 3 weeks whilst participant is on treatment. MTL-CEBPA and pembrolizumab will not be administered on the same day.

Phase 1b of the study will further evaluate safety, tolerability, and assess the clinical activity of MTL-CEBPA and a PD-1 inhibitor (pembrolizumab) in combination.

Participants will receive MTL-CEBPA at a dose considered most appropriate, with regards to safety, tolerability, and efficacy, for further development (based on data from Phase 1a of the study).

Patients with the following (but not limited to) solid tumours will be specifically targeted: breast, lung, ovarian, pancreatic, gall bladder, HCC, neuroendocrine, and cholangiocarcinoma.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female ≥ 18 years
2. Histologically or cytologically confirmed diagnosis of any solid tumour
3. Participants with advanced solid tumours who have progressed on standard of care therapy or for whom no standard therapy is available
4. Participants with advanced pancreatic cancer may also be eligible if they are considered by the treating physician to be unsuitable or have chosen not to take chemotherapy treatment.
5. Participants with high grade serous ovarian, fallopian tube and peritoneal ovarian cancer should have been previously treated with a poly adenosine diphosphate ribose polymerase (PARP)inhibitor and should have received no more than 3 prior lines of systemic therapy.
6. Participants who are naïve to a prior treatment with an immune checkpoint inhibitor. Participants with lung cancer, renal cancer, mesothelioma or melanoma who have received prior PD-1/PD-L1 or a CTLA4 inhibitor containing treatment will be eligible if they have experienced objective response to this treatment (as defined by Response Evaluation Criteria in Solid Tumours [RECIST] 1.1) as part of their most recent treatment line and have had progressive disease occurring within 6 months of the last dose of their checkpoint inhibitor containing treatment.
7. Eastern Cooperative Oncology Group (ECOG)Performance Score0 or 1
8. Life expectancy greater than 3 months at the time of recruitment
9. Measurable disease as per RECIST 1.1 (Response Assessment in Neuro-Oncology [RANO]for glioblastoma multiforme [GBM]) as assessed by the investigator. Lesions situated in a previously irradiated area are considered measurable if progression hasbeen demonstrated in such lesions.
10. In Part 1b of the study, at least one lesion suitable for biopsy (with the exception of brain tumours). If participants have only 1 measurable lesion per RECIST 1.1, the biopsy specimen should be obtained from a non-target lesion.
11. Haematology and clotting profile at screening with no clinically significant findings:

    * Platelet count > 70 x 109/L
    * Absolute neutrophil count ≥ 1.5 x 109/dl

      -≥ 9.0 Serum albumin ≥ 26 g/Lg/dL
    * International Normalised Ratio (INR) < 1.5
12. Adequate renal and hepatic function:

    * Serum albumin ≥ 26 g/L
    * ALT and AST ≤ 2.5x ULN (≤5 × ULN forparticipants with liver metastases and biliary tract cancer)
    * Bilirubin ≤ 1.5 x ULN
    * INR≤ 1.5 x ULN
    * Serum creatinine ≤ 1.5 x ULN
    * Calculated creatinine clearance ≥ 40 mL/min (Cockcroft & Gault). Glomerular filtration rate (GFR) can be used instead of creatinine clearance.
13. Negative blood pregnancy test for women of childbearing potential following a menstrual period (within 10 days prior to first drug administration)
14. For female participants of child-bearing potential, a willingness to use highly effective* contraceptive measures adequate to prevent a new pregnancy for the duration of the study, for at least 6 months after the last dose of MTL-CEBPA or 6 months after the last dose of pembrolizumab, whichever is longer. For women with reproductive potential who use a hormonal method of contraception, concurrent use of a second (barrier) method is recommended.

    *Highly effective methods of birth control are defined as those that result in a low failure rate (i.e., less than 1% per year) when used consistently and correctly (e.g., implants, injectables, oral contraceptives, some intrauterine devices, bilateral tubal occlusion, true sexual abstinence in line with the preferred and usual lifestyle of the participant, or vasectomised partner). For EU countries in particular, see additional requirements in: https://www.hma.eu/fileadmin/dateien/Human_Medicines/01-About_HMA/Working_Groups/CTFG/2014_09_HMA_CTFG_Contraception.pdf Male participants with partners of child-bearing potential are required to use barrier contraception plus an additional contraceptive method that together result in a failure rate of <1% per year during the treatment period and for at least 3 months after the last dose of MTL-CEBPA or 4 months after the last dose of pembrolizumab, whichever is longer. Male participants will also be advised to abstain from sexual intercourse with pregnant or lactating women, or to use condoms. Abstinence is only acceptable if it is in line with the preferred and usual lifestyle of the participant. Periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods), declaration of abstinence for the duration of exposure to investigational medicinal product (IMP), and withdrawal are not acceptable methods of contraception.

    •Note: a woman is considered of child-bearing potential following menarche and until becoming post-menopausal unless permanently sterile. Permanent methods of sterilisation include hysterectomy, bilateral salpingectomy and bilateral oophorectomy. A post-menopausal state is defined as no menses for 12 months without an alternative medical cause(For EU countries in particular please refer to: www.hma.eu/fileadmin/dateien/Human_Medicines/01-About_HMA/Working_Groups/CTFG/2014_09_HMA_CTFG_Contraception.pdf)
15. Able to comply with all the requirements of the protocol.

Exclusion Criteria:

1. Participants who received any prior systemic anticancer therapy investigational drug(s)including vaccines,within the last 30 days prior to study treatment initiation (Cycle1 Day 1)
2. Grade > 1 prior treatment-related toxicity at the time of screening, with the exception of alopecia or Grade 2 neuropathy which may be eligible if recovered tobaseline and upon discussion with the Sponsor.
3. Participants received prior radiotherapy within 2 weeks of start of study treatment
4. Participants not recovered adequately from major surgery or radiotherapy.
5. Participants with history of clinically significant haemorrhage or gastrointestinal perforation•Participants with history of bilateral portal vein occlusion
6. Known infection with human immunodeficiency virus (HIV)withCD4+ T-cell counts <350 cells/μL or with a history of acquired immune deficiency syndrome (AIDS)-defining opportunistic infection
7. Participants with known history of infection with hepatitis B(HBV)(defined as hepatitis B surface antigen [HBsAg] reactive) or known infection with hepatitis C (defined as detectable HCV RNA via qualitative nucleic acid testing). Note -this exclusion criterion does not apply to participants with HCC. For participants with HCC only: participants with past or ongoing HCV infection will be eligible for the study but must have completed their treatment at least 1 month prior to starting study intervention and their HCV viral load has to be below the limit of quantification. Participants who are HCV antibody (HCVAb positive but HCV RNA negative, due to prior treatment or natural resolution, will be eligible. Participants with past or controlled ongoing HBV will be eligible as long as their HBV viral load is less than 500 IU/mL prior to first dose of study drug. Participants on active HBV therapy with viral loads under 100 IU/mL should stay on the same therapy throughout study intervention.
8. Symptomatic, untreated, or actively progressing central nervous system (CNS) metastases and/or carcinomatous meningitis, with the exception of participants with GBM. Participants with previously treated metastases may participate provided they are radiologically stable for at least 4 weeks by repeat imaging performed during study screening, clinically stable, and without requirement for steroid treatment above 10mg/day (prednisone) for at least 28days prior to the first dose of study intervention. An MRI brain scan for all participants with stable brain metastases at screening (CT scan will be allowed if MRI is contraindicated).
9. Participants with clinically significant, progressing malignant ascites except for those with ovarian tumours•Participants with known history of non-infectious pneumonitis, myocarditis, or nephritis•Signs and symptoms of heart failure within the last 12 months characterised as greater than New York Heart Association (NYHA) Class I or other clinically significant cardiac abnormalities (such as myocardial infarction) including stable abnormalities.
10. Major surgery within the last 30 days prior to study treatment initiation. Participants must have recovered adequately from the procedure and/or any complications from the surgery prior to starting study intervention.
11. Participants with history of solid organ or haematological transplantation•Participants with sepsis, ineffective biliary drainage with or without cholangitis, obstructive jaundice or encephalopathy at screening visit or within the last 2weeks prior to study treatment initiation, whichever is earlier
12. Evidence of spontaneous bacterial peritonitis or renal failure, or allergic reaction at screening visit or within the last 2 weeks prior to study treatment initiation, whichever is earlier•Pregnant or lactating women
13. Received systemic corticosteroids and other immunosuppressants in the 4 weeks prior to enrolment into the study (please see note on exception details in Section 6.3.1).
14. Received live (attenuated) vaccine in the 30 days prior to first dose of study drug.Live vaccines include, but are not limited to: measles, mumps, rubella, varicella/zoster chicken pox), yellow fever, rabies, Bacillus Calmette-Guérin (BCG), and typhoid vaccine. Seasonal influenza and COVID-19 vaccines for injection are generally inactive/not viablevirus vaccines and are allowed; however, intranasal influenza vaccines (e.g., FluMist®) are live attenuated vaccines and are not allowed.
15. Active or prior documented autoimmune or inflammatory disorders (including inflammatory bowel disease [e.g., colitis or Crohn's disease]requiring immunosuppressive treatment, diverticulitis [with the exception of diverticulosis], systemic lupus erythematosus, Sarcoidosis syndrome, or Wegener syndrome [granulomatosis with polyangiitis, Graves' disease, rheumatoid arthritis, hypophysitis, uveitis, etc]). The following are exceptions to this criterion:

    * Participants with vitiligo or alopecia.
    * Participants with hypothyroidism (e.g., following Hashimoto syndrome) euthyroid on hormone replacement.
    * Any chronic skin condition that does not require systemic therapy.
    * Participants without active disease in the last 2 years may be included but only after consultation with the study physician.
    * Participants with coeliac disease controlled by diet alone.
16. Participants with an active infection requiring systemic therapy.
17. Known hypersensitivity to the active substance (pembrolizumab) or to any of the excipients.
18. Any known additional malignancy requiring active treatment within the past 3 years. Exceptions include early-stage cancers such carcinoma in situ or stage 1, such as melanoma, basal cell carcinoma or squamous cell carcinoma of the skin, in situ cervical cancer, or in situbreast cancer, which have been treated with curative intent.
19. Any other condition (including psychiatric or substance abuse, known or suspected poor compliance, etc.), therapy, or laboratory finding that, in the judgement of the investigator, may affect the participant's ability to participate, fully follow the protocol specific procedures, or is not in the best interest of the participant to take part in the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2019-11-13 (Actual); Primary Completion 2025-01-25 (Actual); Study Completion 2025-01-25 (Actual)

PRIMARY OUTCOMES:
Adverse events | From screening visit through study completion, an average of 1 year
  Frequency of adverse events graded according to toxicity criteria (NCI CTCAE v 5.0) and categorised by body system and diagnosis.
Anti-tumour activity | information on how the event is determined and over what estimated period of time (e.g., "From date of sceening visit until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 60 months
  Change from baseline CT scan using the revised Response Evaluation Criteria in Solid Tumours (RECIST) guideline version 1.1 modified RECIST(mRECIST) and irRECIST

SECONDARY OUTCOMES:
Pharmokinetic analysis of the study drug MTL-CEBPA when co administered with pembrolizumab | Blood samples will be collected on Days 1, 2, 3, 4, 8, 9 10, and 11 of the study
  Blood sampling Blood samples collected at pre-defined timepoints will be analysed to define the maximum plasma concentration (Cmax) of MTL-CEBPA after intravenous administration.

CONTACTS AND LOCATIONS:
Overall Officials: Nagy Habib, ChM, FRCS, Study Director — Mina Alpha Limited
Locations (3):
- United Kingdom (3):
  - Guys and St Thomas NHS Foundation Trust, London
  - Imperial College Healthcare NHS Trust, London
  - Freeman Hospital, Newcastle Upn Tyne Hospitals NHS Foundation Trust, Newcastle upon Tyne

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Plummer R, Sodergren MH, Hodgson R, Ryan BM, Raulf N, Nicholls JP, Reebye V, Voutila J, Sinigaglia L, Meyer T, Pinato DJ, Sarker D, Basu B, Blagden S, Cook N, Jeffrey Evans TR, Yachnin J, Chee CE, Li D, El-Khoueiry A, Diab M, Huang KW, Pai M, Spalding D, Talbot T, Noel MS, Keenan B, Mahalingam D, Song MS, Grosso M, Arnaud D, Auguste A, Zacharoulis D, Storkholm J, McNeish I, Habib R, Rossi JJ, Habib NA. TIMEPOINT, a phase 1 study combining MTL-CEBPA with pembrolizumab, supports the immunomodulatory effect of MTL-CEBPA in solid tumors. Cell Rep Med. 2025 Apr 15;6(4):102041. doi: 10.1016/j.xcrm.2025.102041. Epub 2025 Mar 31. PMID 40168999
- [Derived] Hashimoto A, Sarker D, Reebye V, Jarvis S, Sodergren MH, Kossenkov A, Sanseviero E, Raulf N, Vasara J, Andrikakou P, Meyer T, Huang KW, Plummer R, Chee CE, Spalding D, Pai M, Khan S, Pinato DJ, Sharma R, Basu B, Palmer D, Ma YT, Evans J, Habib R, Martirosyan A, Elasri N, Reynaud A, Rossi JJ, Cobbold M, Habib NA, Gabrilovich DI. Upregulation of C/EBPalpha Inhibits Suppressive Activity of Myeloid Cells and Potentiates Antitumor Response in Mice and Patients with Cancer. Clin Cancer Res. 2021 Nov 1;27(21):5961-5978. doi: 10.1158/1078-0432.CCR-21-0986. Epub 2021 Aug 18. PMID 34407972
- See also: Company web page — http://www.minatx.com